CLINICAL TRIAL: NCT00130260
Title: Phase 3b Multicenter, Randomized, Placebo-Controlled, Double-Blind Study Evaluating Immunogenicity and Safety of a 3rd and 4th Dose of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine in Adults With End-Stage Renal Disease
Brief Title: Evaluation of a Third and Fourth Dose of StaphVAX® in Adults With End-Stage Renal Disease
Acronym: SHIELD-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: unsatisfactory efficacy data from preceding trial
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Matt Hohenboken, MD, PhD, Executive Director Clinical & Medical Affairs, Nabi Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nabi-1372
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Staphylococcal Infections; Chronic Kidney Failure
Keywords: Staphylococcus aureus; Vaccine; Randomized Controlled Trial
MeSH Terms: conditions — Staphylococcal Infections; Kidney Failure, Chronic | interventions — StaphVax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- vaccine, schedule 1 (Experimental): 3rd and 4th dose of vaccine, on original schedule
  Interventions: Biological: Staph aureus types 5 and 8 conjugate vaccine
- vaccine, schedule 2 (Experimental): 3rd and 4th dose of vaccine on modified schedule
  Interventions: Biological: Staph aureus types 5 and 8 conjugate vaccine
- placebo, schedule 1 (Placebo Comparator): 3rd and 4th dose of placebo, on original schedule
  Interventions: Biological: placebo
- placebo, schedule 2 (Placebo Comparator): 3rd and 4th dose of placebo on modified schedule
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Staph aureus types 5 and 8 conjugate vaccine — each IM dose contains 200 mc total conjugate
  Other Names: StaphVAX®
  Arms: vaccine, schedule 1; vaccine, schedule 2
Biological: placebo — placebo to match StaphVAX
  Arms: placebo, schedule 1; placebo, schedule 2

SUMMARY:
This study is a continued evaluation of the immune response to StaphVAX , a Staphylococcus aureus type 5 and 8 capsular polysaccharide conjugate vaccine, in end-stage renal disease patients, by giving a 3rd and 4th dose to a subset of the participants in the previous efficacy trial. Participants continue to receive the vaccine or placebo in a blinded manner, and are also randomly assigned to 1 of 2 different intervals between the doses. The immunogenicity is measured by the antibodies in the blood, and typical vaccine safety information is also collected.

ELIGIBILITY:
Inclusion Criteria:

* Participation in prior study Nabi-1371
* Written informed consent
* Negative serum pregnancy test, where appropriate
* Expect to comply with protocol procedures and schedule

Exclusion Criteria:

* Known HIV
* Immunomodulatory drugs
* Malignancy (other than basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or early stage prostate cancer)
* Active infection in the 2 weeks prior to study injection
* Serious S. aureus infection within the last 2 months prior to injection
* Hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-08; Primary Completion 2005-12 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
serotype-specific antibody concentrations | 6 weeks after each dose

SECONDARY OUTCOMES:
serotype-specific antibody concentrations | at several other time points up to 12 months after dose
elicited vaccine reactogenicity | daily for 7 days after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- multiple sites: contact Central Study coordination, Birmingham, Alabama, United States